CLINICAL TRIAL: NCT00335413
Title: Autoregulation of Glomerular Filtration Rate in Patients With Type 1 Diabetes During Spironolactone Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2006-001453-10; 2612-3144; KA-20060055
Record Dates: First submitted 2006-06-07; First posted 2006-06-09 (Estimated); Last update posted 2008-06-05 (Estimated); Status verified 2008-06

CONDITIONS: Hypertension
Keywords: Renal autoregulation; Glomerular filtration rate; Type 1 diabetes
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 1 | interventions — Spironolactone

INTERVENTIONS:
Drug: Spironolactone

SUMMARY:
To evaluate the impact of spironolactone treatment on renal autoregulation in hypertensive type 1 diabetic patients.

DETAILED DESCRIPTION:
Double-masked, randomized, crossover trial. In random order, patients will be treated with spironolactone 25 mg o.d. and matched placebo for 28 days.

On the last day of treatment, GFR will be determined twice on the same day: first without clonidine and secondly after injection of clonidine (clonidine induces a transient reduction in blood pressure, with no influence on renal plasma flow and GFR), in order to evaluate the effect of antihypertensive treatment with spironolactone on renal autoregulation of GFR.

The study will be preceded by a wash-out period of 1 month for patients receiving antihypertensive medication. Patients will be instructed to measure blood pressure twice daily, three days a week during this period. If, during the washout period, blood pressure exceeds 170/105 mm Hg or persistent edemas develop, treatment with long-acting loop diuretics will be initiated and continued throughout the rest of the study. If blood pressure despite diuretic treatment still exceeds 170 mm Hg systolic and/or 105 mm Hg diastolic, the patient will be excluded from the study and previous/appropriate antihypertensive treatment will be restarted.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Age between 18 and 70 years
* Blood pressure ≥ 135 mm Hg systolic and/or ≥ 85 mm Hg diastolic or ongoing antihypertensive treatment
* Informed consent

Exclusion Criteria:

* Diabetic nephropathy
* Other known kidney or renal tract disease
* Malignant hypertension
* Blood pressure > 170/105 at baseline or during AHT wash-out period
* Plasma potassium > 4.7 mmol/l
* Elevated plasma creatinine (>88 µmol/l for women and >100 µmol/l for men)
* Symptoms of Ischemic heart disease within 3 months prior to study start
* Previous cerebrovascular event (apoplexy, TCI)
* Abuse of medicine or alcohol
* Pregnancy or breastfeeding
* Woman of child-bearing age who are not using adequate contraception
* ASA treatment > 1g/day or regular use of NSAIDs
* Known allergy to or side-effects of spironolactone
* Inability to understand patient information

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2006-06; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Changes in glomerular filtration rate

SECONDARY OUTCOMES:
Changes in blood pressure
Changes in albuminuria
Changes in fractional albumin clearance

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Henrik Parving, MD,DMSc,Prof, Principal Investigator — Steno Diabetes Center Copenhagen

REFERENCES:
- [Derived] Chung EY, Ruospo M, Natale P, Bolignano D, Navaneethan SD, Palmer SC, Strippoli GF. Aldosterone antagonists in addition to renin angiotensin system antagonists for preventing the progression of chronic kidney disease. Cochrane Database Syst Rev. 2020 Oct 27;10(10):CD007004. doi: 10.1002/14651858.CD007004.pub4. PMID 33107592